CLINICAL TRIAL: NCT04455048
Title: The Effectiveness of Manipulation Treatment in Acute Cervical Region Pain
Brief Title: The Effectiveness of Manipulation Treatment in Cervical Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-RK-04
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain
Keywords: Tape; Pain; Rehabilitation
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Intervention Model Description: Two groups with a sham control. Assessments will be performed before manipulation, immediately after first session, in the second week, and two months after the last session.
Who Masked: Participant, Outcomes Assessor
Masking Description: The manipulation group will receive a single session thrust manipulation and the control group will receive a sham manipulation. Outcome assessment will be performed by another investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A single-session manipulation with a high-speed low-amplitude thrust technique in the cervicothoracic transition region will be applied each week for two weeks.
  Interventions: Other: Cervicothoracic thrust manipulation
- Control Group (Sham Comparator): A sham manipulation without a high-speed low-amplitude thrust technique in the cervicothoracic transition region will be applied.
  Interventions: Other: Cervicothoracic thrust manipulation sham

INTERVENTIONS:
Other: Cervicothoracic thrust manipulation — The patient will be positioned in a supine position with arms crossed over over the trunk and holding the shoulders. The therapist will place a stabilizing hand over transverse process of T1 in pistol grip and contacted patients elbow with sternum and patient will be asked do a hip bridge while taking a deep breath than exhale. Thrust manipulation will be applied at the end of exhale.
  Arms: Intervention Group
Other: Cervicothoracic thrust manipulation sham — The patient will be positioned in a supine position with arms crossed over over the trunk and holding the shoulders. The therapist will place a stabilizing hand over transverse process of T1 in pistol grip and contacted patients elbow with sternum and patient will be asked do a hip bridge while taking a deep breath than exhale. A soft compression will be applied at the end of exhale without a thrust.
  Arms: Control Group

SUMMARY:
Neck pain is the second most common musculoskeletal pain after lumbar pain. Prevalence is 27.2% female and 17.4% in male population (1, 2). Approximately 1/3 of acute onset neck aches become chronic. It causes increasing the cost of treatment and also the loss of labor (3, 4).

DETAILED DESCRIPTION:
Acute neck pain is often caused by mechanical causes and can be classified as rheumatic diseases, infectious and tumoral pathologies, metabolic bone diseases such as osteoporosis and osteomalacia, pain reflected the cervical region. A-V malformation and syringomyelia are the causes of chronic cervical pain (5). Mechanical neck pain is a non-radicular pain caused by local musculoskeletal structures and is characterized by a spasm of the cervical muscles. (6, 7). Posture, emotional stress, cold and fatigue are etiologic causes, and pain is also reflected in the cervical, occipital and scapular regions depending on the severity of muscle spasm and the presence of trigger point in myofascial pain syndrome (9, 10). Many authors have suggested that facet joints are associated with mechanical dysfunction as a common cause of cervical pain (8-10).

The pain in the head and neck region affects the quality of life, cognitive and functional status of the person. The most important difficulty and failure in the treatment of such pain arise from the inability to diagnose the disease correctly. Good anatomical and biomechanical properties of the region, comprehensive anamnesis, physical examination under static and dynamic conditions, laboratory and radiological examinations are the most important milestones of diagnosis (12). In most cases, medical treatment and physical therapy modalities (superficial and deep heat, electrotherapy, laser, traction, massage, spa) are sufficient for pain relief and recovery of function, but interventional procedures and surgical procedures are needed for the fewer patient. Recently, spinal mobilization and manipulation techniques can be used to relieve pain and restore function in the early stages. Although it is a safe method, in order to prevent the rare complications it is necessary to determine the indications of treatment correctly, to exclude contiguous cases and to apply the manipulation by experts (12).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis Nonspecific neck pain (NSNP)
* Symptoms should last longer than 2 weeks

Exclusion Criteria:

* Any known cause such as radiculopathy or neurological diseases,
* History of neck surgery,
* History of vertebral fracture,
* Osteoporosis,
* Tumor or a mass in the vertebral column,
* Any spinal thrust manipulation contraindication,
* Medication usage such as antiinflammatory or analgesic which might effect outcome assessments,
* History of spinal manipulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | two weeks
  Pain pressure threshold (PPT). was assessed with an analogue algometry (Baseline, FEl Inc. White Plains, NY,USA) with 1 cm2 rubber tip was used to measure the pain pressure threshold. Algometer perpendicularly placed over spinous process of T1 on prone position and pressure progressively increased 1 kg/s until patients verbally reported pain under the tip of algometer or referring pain. Measurement repeated three times and average score recorded.

SECONDARY OUTCOMES:
Visual analog scale | two weeks
  The patient was asked to mark the severity of his or her pain with active motion on a horizontal line 100 millimeters in length. The intensity of the pain was calculated by measuring the area in which the individual marked between 0 (no pain) and 10 (the most severe pain I felt in my life).
Cervical range of motion | two weeks
  Cervical Range of Motion (ROM) of flexion,extension, lateral flexion and rotation were measured with basic cervical ROM device (Performance Attainment, Associates, St Paul, MN, USA) in seated position without back support.
Neck Disability Index | two weeks
  Perceived disability of patients was assessed with 10-item item Neck Disability Index (NDI),which a modified from Oswestry Low Back Pain Disability Index to assess with a score range of 0 to 50.
Global Perceived Effect Scale | two weeks
  Change in the perception of the symptoms after the treatment was measured by a Global Perceived Effect Scale. Patients were asked to rate change between 1 completely recovered, 4 unchanged, 7 vastly worse on a horizontal likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Erdal Dilekçi, MD, Principal Investigator — Bolu Abant Izzet Baylsa University; Ramazan KURUL, Ph.D, Principal Investigator — Bolu Abant Izzet Baylsa University
Locations (2):
- Turkey (Türkiye) (2):
  - Abant Izzet Baysal University, Bolu, Merkez
  - Health Sciences Faculty Bolu Abant Izzet Baysal University, Bolu, Merkez

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after study publicaiton with online link.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after study published and will be available indefinetly.
Access Criteria: data will be accessed from cloud store link